CLINICAL TRIAL: NCT06125470
Title: Healthy Families for Pakistan Through Accelerating Gender-responsive Sexual Reproductive Health (SRH) and Family Planning (FP) Services
Brief Title: SihatMand Khandaan Healthy Families for Pakistan
Acronym: SMK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Global Affairs Canada (Other); United Nations (Other)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Distinguished University Professor, Aga Khan University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-3606-11051
Record Dates: First submitted 2021-08-31; First posted 2023-11-09 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Contraception; Contraception Behavior; Reproductive Behavior; Maternal Behavior
MeSH Terms: conditions — Contraception Behavior; Reproductive Behavior | interventions — Private Sector; Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: Strengthened technical capacity of healthcare workforce to provide quality gender-responsive SRH /FP services to women of reproductive age, youth and adolescents. .
  Increased availability of quality gender-responsive materials, equipment and appropriate infrastructure for FP/SRH Enhanced ability of district and provincial health authorities to maintain adequate and sustainable supplies of FP commodities Improved knowledge and attitudes regarding FP/SRH amongst male and female community members Enhanced ability of local community structures, institutions and leaders to identify and respond to gender and social barriers to utilization of FP/SRH services.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention areas (Experimental): Health facilities and other service delivery points including outreach health workers receiving FP supplies, trainings and renovations to create enabling environment at health and Family planning facilities Community engagement and creating creating adolescents friendly spaces roll out of Gender responsive strategies
  Interventions: Behavioral: Uptake of quality Reproductive health and Family planning products, information and Services; Behavioral: Capacity building of facility based and community based healthcare providers (public and private sector) on FP /SRH; Behavioral: Adolescent Engagement; Behavioral: Renovation and Refurbishment of selected healthcare facilities; Behavioral: Use of Data for Effective Decision-making; Behavioral: Procurement of FP/SRH medical supplies and equipment

INTERVENTIONS:
Behavioral: Uptake of quality Reproductive health and Family planning products, information and Services — Strengthening capacity of health facilities and outreach to deliver quality reproductive and family planning services and address demand side barriers to the uptake of the services
Behavioral: Capacity building of facility based and community based healthcare providers (public and private sector) on FP /SRH — Training sessions on FP / SRH including FP Methods - LARC, PPIUD - Task Sharing & Shifting for facility based healthcare providers at provincial level for Master Trainers with trickle down sessions at district level.
  Training on Sayana Press, ECP, Balance Counselling Strategy and Life Skills Based Education for community-based healthcare providers including LHWs at district level.
Behavioral: Adolescent Engagement — Identification of adolescent-friendly spaces through community based platforms including LHW health houses for girls and village health committees for boys with context-appropriate arrangements for LSBE and SRH counselling.
Behavioral: Renovation and Refurbishment of selected healthcare facilities — Identification and improvement/ renovation of public and private healthcare facilities to strengthen the quality, provision and delivery of FP/SRH services, especially counselling, to catchment population
Behavioral: Use of Data for Effective Decision-making — Improvement in data recording at the source level with reporting at existing platforms i.e. DHIS and LHW-MIS and use of this data for local decision making
Behavioral: Procurement of FP/SRH medical supplies and equipment — Provision of commodities / supplies for shortest-time possible in facilities having stock-outs

SUMMARY:
The SMK project's primary goal is to improve the status of SRH of women and adolescents within those targeted areas which feature inadequate progress on existing SRH indicators. The focus remains on empowering increasingly marginalized and vulnerable populations to exercise their reproductive rights, free of coercion, discrimination and violence. This will be achieved through the implementation of evidence-based and socio-culturally sensitive FP/ SRH interventions within ten districts of Pakistan. The aim of this project is therefore to evaluate the impact of a package of community and facility-based interventions on improving the SRH/ FP of the targeted population.

In order to achieves this, a quasi-experimental pre & post evaluation intervention study with a formative phase, baseline assessment, intervention phase and finally an end-line assessment, consisting of both qualitative & quantitative monitoring & evaluation tools will be applied at the household, community, healthcare facility and district levels in all project areas.

Furthermore, descriptive statistics will be tabulated on key indicators and stratified on selected variables. Means for continuous variables and proportion for categorical variables will be calculated at a 95% confidence interval within this study

DETAILED DESCRIPTION:
A Quasi experimental pre & post evaluation intervention study with a formative research design will be adopted. This study will have three phases; (i) pre-assessment (baseline assessment, quantitative assessment & qualitative assessment - FGDs & In-depth Interviews), (ii) intervention and (iii) post assessment. The pre and post assessment will employ a mixed methodology approach.

The primary purpose of the pre-evaluation is to identify the FP / SRH related needs of the targeted population and existing gaps in health service delivery. These will effectively inform the interventions to be implemented. The post-evaluation will encompass mechanisms for quality assurance and monitoring of project impact and sustainability. Both pre and post- evaluations will be conducted using the same tools.

The overarching objective is therefore to evaluate the impact of a package of community and facility-based interventions on the SRH of the targeted population as delivered through the specific objectives outlined below:

1. To roll out effective, gender-responsive and COVID-19 appropriate interventions related to maternal, reproductive and newborn health in the public and private sector for the selected districts in the three provinces of Pakistan.
2. To generate data on knowledge, attitude, practices, access and use of health services for the selected districts.
3. To identify areas for capacity building and training for healthcare providers to improve quality and delivery of FP /SRH (as affected by the ongoing COVID-19 pandemic) for the selected districts.
4. To understand and explore the gender and social barriers to utilization and uptake of FP /SRH services by members of the community within the selected districts.

ELIGIBILITY:
Inclusion Criteria:

* Married women of reproductive age living in the project areas

Exclusion Criteria:

* Not residing in the area for more than six months

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 236000 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Contraceptive Prevalence Rate | over the period of 3 years
  Contraceptive prevalence is the percentage of women who are currently using, or whose sexual partner is currently using, at least one method of contraception, regardless of the method used. It is usually reported for married or in-union women aged 15 to 49.

SECONDARY OUTCOMES:
Unmeet need for Family planning | over the period of 3 years
  Women with unmet need are those who are fecund and sexually active but are not using any method of contraception, and report not wanting any more children or wanting to delay the next child. The concept of unmet need points to the gap between women's reproductive intentions and their contraceptive behaviour.
Skilled birth rate | over the period of 3 years
  A birth attendant, also known as skilled birth attendant, is a health professional who provides basic and emergency care to women and their newborns during pregnancy, childbirth and the postpartum period.
Antenatal coverage | over the period of 3 years
  at least one visit to skilled birth attendant during pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No